CLINICAL TRIAL: NCT02352311
Title: A Randomized, Open-label, Single-dose, 2-treatment, 2-way, 2-period Crossover Study to Evaluate the Safety and the Pharmacokinetic Characteristics of DKF-313 in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetic Characteristics of DKF-313
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DK-DT-002
Record Dates: First submitted 2015-01-22; First posted 2015-02-02 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2015-02

CONDITIONS: Benign Prostate Hyperplasia; Healthy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 AVODART, CIALIS, DKF-313 (Experimental): In Period 1, AVODART (dutasteride) soft gelatin capsule and CIALIS (tadalafil) tablet 5 mg are administered as single dose. In Period 2, DKF-313 tablet (dutasteride 0.5 mg and tadalafil 5 mg) is administered as single dose.
  Interventions: Drug: DKF-313; Drug: AVODART; Drug: CIALIS
- Arm 2 DKF-313, AVODART, CIALIS (Experimental): In Period 1, DKF-313 tablet (dutasteride 0.5 mg and tadalafil 5 mg) is administered as single dose. In Period 2, AVODART (dutasteride) soft gelatin capsule and CIALIS (tadalafil) tablet 5 mg are administered as single dose.
  Interventions: Drug: DKF-313; Drug: AVODART; Drug: CIALIS

INTERVENTIONS:
Drug: DKF-313 — Combination of dutasteride 0.5 mg and tadalafil 5 mg
Drug: AVODART — Dutasteride 0.5 mg
  Other Names: Dutasteride
Drug: CIALIS — Tadalafil 5 mg
  Other Names: Tadalafil

SUMMARY:
This is a randomized, open-label, single-dose, 2-treatment, 2-way, 2-period crossover study to evaluate the safety and the pharmacokinetic characteristics of DKF-313 (dutasteride and tadalafil) in healthy male volunteers.

DETAILED DESCRIPTION:
This study is conducted to evaluate the pharmacokinetics of DKF-313 (dutasteride and tadalafil) comparing with the concomitant administration of AVODART and CIALIS in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 to 29 years
2. BMI 17.5 to 30.5 kg/m2 and body weight 55 kg or more
3. No congenital or chronic diseases within 3 years, no disease symptoms or findings
4. Eligible according to the laboratory results of hematology, blood chemistry and urinalysis and ECG
5. Voluntarily signed the informed consent form 6. Willing to participate in the study

Exclusion Criteria:

1. Clinically significant disorders of blood, kidney, endocrine, respiratory system, gastrointestinal system, urology, cardiovascular system, liver, psychiatry, neurology or allergy
2. Gastrointestinal diseases or surgery which may affect absorption of the investigational products
3. ALT or AST > 2xULN
4. Excessive alcohol consumption (> 210 g/week) within 6 months
5. Participated and administered the investigational products in other clinical trial within 2 months
6. SBP ≤ 100 mmHg or ≥ 150 mmHg or DBP ≤ 60 mmHg or ≥ 100 mmHg
7. History or positive result of serious alcohol or drug abuse within 1 year
8. Drugs which induce or inhibit drug metabolism within 1 month
9. Smoked more than 10 cigarettes a day
10. Prescribed drugs or over-the counter drugs within 10 days
11. Donated whole blood within 2 months or apheresis within 1 month
12. Severe acute/chronic medical and mental conditions or lab abnormalities which may increase the risk or interfere in the interpretation of study results
13. Hypersensitivity to tadalafil or phosphodiesterase type 5 inhibitor, and dutasteride or 5-α reductase inhibitor, or other drugs including aspirin, antibiotics, etc.
14. Galactose intolerance, fructose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
15. CYP3A4 inhibitors or CYP3A4 inducers within 2 weeks
16. Myocardial infarction within 90 days
17. Unstable angina or angina during sexual intercourse
18. Heart failure (New York Heart Association Class 2 or higher) within 6 months
19. Uncontrolled arrhythmias
20. Stroke within 6 months
21. Inherited retinal degeneration including retinitis pigmentosa
22. Vision loss in one eye due to non-arteritic anterior ischemic optic neuropathy (NAION)
23. Plans to donate blood for at least 6 months after final dose of the investigational products
24. Unwilling to comply with the lifestyle guidelines in the protocol
25. Not eligible due to other reasons at the investigator's discretion

Ages: 19 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
AUClast and Cmax of dutasteride and tadalafil | 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 144, 192 h

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, M.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea